CLINICAL TRIAL: NCT04227301
Title: Influence of Serum Sodium Levels on Bone Metabolism and Turnover in Hospitalized Patients - A Prospective Study (BONA-Trial)
Brief Title: Influence of Serum Sodium Levels on Bone Metabolism and Turnover in Hospitalized Patients
Acronym: BONA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01858; me18ChristCrain6
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hyponatremia
Keywords: electrolyte disorder; Bone Metabolism; Sodium Levels
MeSH Terms: conditions — Hyponatremia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological material, i.e. blood samples, will be handled according to good clinical practice and good laboratory practice. Samples will be collected in secure containers (Sarstedt Monovette®) and will be centrifuged to collect serum. Serum will be stored at - 70°C in a thermo-controlled ultra-deep freezer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyponatremic patients: Patients hospitalized at the University Hospital of Basel and presenting with hyponatremia will be screened for the study
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling for measurement of bone markers after a fasting period of at least 6 hours

SUMMARY:
In this study, the possible role of serum sodium concentration and its changes on bone markers in hospitalized, hyponatremic patients is determined. Therefore, it is investigated whether in hospitalized, hyponatremic patients the level of carboxy-terminal collagen crosslinks (CTX) is modified by changes in plasma sodium concentration, independently from the aetiology of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Adult hospitalized patients with non-hypertonic hyponatremia: serum sodium < 130 mmol/l, serum osmolality < 300 milliosmol /kg
* age 18 to 99-year-old
* Informed consent as documented by signature

Exclusion Criteria:

* Severe symptomatic hyponatremia in need of intensive care treatment
* Hypertonic hyponatremia with serum osmolality > 300 mOsm/kg
* End of life care (palliative treatment)
* End stage kidney disease (dialysis)
* Acute liver failure
* Wernicke encephalopathy
* Hepatic encephalopathy during last 2 months
* Hepato-renal syndrome
* Any bone disease requiring treatment in the last three years
* History of fragility fractures
* Pre-menopausal women
* Hypogonadism (diagnosed before hospitalization)
* Hyperthyroidism
* Steroid therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients (18 to 99-year-old), with non-hypertonic hyponatremia
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change in carboxy-terminal collagen crosslinks (CTX) levels | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  CTX level (pg/ml) and its dynamic within 10 days of hospitalization
Change in plasma sodium level | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  serum sodium levels (milliequivalents per liter (mEq/L) and its dynamic within 10 days of hospitalization

SECONDARY OUTCOMES:
Changes in bone specific alkaline phosphatase (bAP) | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  bAP levels and their dynamic within 10 days of hospitalization
Change in osteocalcin | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  Osteocalcin (ng/mL) levels and their dynamic within 10 days of hospitalization
Change in procollagen type I N propeptide (PINP) (PINP) levels | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  PINP (ng/mL) levels and their dynamic within 10 days of hospitalization
Change in sclerostin | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  Sclerostin (pg/ml) levels and their dynamic within 10 days of hospitalization
Change in parathyroid hormone (PTH) | changes from baseline (day 1) to day 10 after inclusion in the study
  PTH (pg/ml) levels and their dynamic within 10 days of hospitalization
Change in 25-hydroxy-vitamin D3 | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  25-hydroxy-vitamin D3 (ng/ml) levels and their dynamic within 10 days of hospitalization
Change in calcium | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  Calcium (mg/dl) levels and their dynamic within 10 days of hospitalization
Change in phosphate levels | baseline blood exam on day 1 after inclusion and further blood collections at day 10 (+/-3 days) or at discharge, if discharge will be earlier
  Phosphate(mg/dl) levels and their dynamic within 10 days of hospitalization
Numbers of falls | numbers of falls within 30 days after enrolment
  telephone interview will be performed to collect data about occurrence and numbers of falls within 30 days after enrolment
Numbers of fractures | Numbers of fractures within 30 days after inclusion in the study
  telephone interview will be performed to collect data about occurrence and numbers of fractures within 30 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med, Principal Investigator — Endocrinology, Diabetology and Metabolism, University Hospital Basel
Locations (1):
- Endocrinology, Diabetes and Metabolism, University Hospital Basel, Basel, Switzerland